CLINICAL TRIAL: NCT05953428
Title: Reducing Postoperative Opioids in Patients Undergoing Laparoscopic Hiatal Hernia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Steven Greenberg, Jeffery S. Vender Endowed Chair of Anesthesiology Research and Education, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EH23-020
Record Dates: First submitted 2023-07-05; First posted 2023-07-20 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Hiatal Hernia
Keywords: Opioid Sparing Anesthesia Protocol; Opioid Based Anesthesia Protocol
MeSH Terms: conditions — Hernia, Hiatal

STUDY DESIGN:
Intervention Model Description: Patients undergoing laparoscopic hiatal hernia repairs will be randomized to:
  Experimental Group: Opioid Sparing Anesthesia Protocol vs. Control Group: Opioid Based Anesthesia Protocol
Who Masked: Participant, Care Provider
Masking Description: The study participants, surgeons and PACU nurses will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Opioid Sparing Anesthesia Protocol (Experimental): The OSA protocol will include boluses of dexmedetomidine and ketamine at anesthesia induction, followed by a ketamine infusion that will continue until PACU discharge. Another bolus of ketamine will be administered upon surgical incision and another dexmedetomidine bolus will be given at surgical closure to reduce the use of opioids.
  Interventions: Other: Opioid Sparing Anesthesia Protocol (OSA)
- Opioid Based Anesthesia Protocol (Other): The OBA group will be administered a saline infusion at the same rate of the ketamine infusion (only while in the PACU) up until PACU discharge so that surgeons, patients, and PACU nurses will be blinded. The OBA group will be administered fentanyl 100 mcg IV for anesthesia induction followed by 50 mcg IV boluses when heart rate or systolic blood pressure is 20% above baseline throughout the case.
  Interventions: Other: Opioid Based Anesthesia Protocol (OBA)

INTERVENTIONS:
Other: Opioid Sparing Anesthesia Protocol (OSA) — OSA protocol will include boluses of dexmedetomidine and ketamine at anesthesia induction, followed by a ketamine infusion that will continue until PACU discharge. Another bolus of ketamine will be administered upon surgical incision and another dexmedetomidine bolus will be given at surgical closure to reduce the use of opioids.
  Arms: Opioid Sparing Anesthesia Protocol
Other: Opioid Based Anesthesia Protocol (OBA) — The OBA group will be administered a saline infusion at the same rate of the ketamine infusion (only while in the PACU) up until PACU discharge so that surgeons, patients, and PACU nurses will be blinded. The OBA group will be administered fentanyl 100 mcg IV for anesthesia induction followed by 50 mcg IV boluses when heart rate or systolic blood pressure is 20% above baseline throughout the case.
  Arms: Opioid Based Anesthesia Protocol

SUMMARY:
This is a prospective randomized, double-blinded, controlled trial that will enroll 75 subjects undergoing laparoscopic hiatal hernia repair surgery. Participants who meet eligibility criteria will be randomized in a 1:1 ratio to receive either the opioid sparring anesthesia protocol (OSA) or the opioid based anesthesia protocol (OBA). The purpose of this study is to investigate if an opioid sparring protocol for laparoscopic hiatal hernia repair will reduce opioid consumption during discharge. Other outcomes include: postoperative VAS scores (PACU arrival, PACU discharge, hospital discharge), total in hospital opioid consumption, PACU length of stay, incidence of postoperative nausea and vomiting (PONV in PACU, postoperative day 1, during hospital stay), rehospitalization rate, rate of reoperation, rate of emergency room visit, surgeon satisfaction, and hospital cost differential.

DETAILED DESCRIPTION:
The administration of perioperative opioids to nearly 80% of surgical patients leaves approximately 6 million Americans susceptible to becoming opioid-dependent. This practice has been hypothesized as a contributing factor to the ongoing opioid crisis, where currently more than 136 Americans die from an opioid overdose every day. Recent data suggest a potential benefit of reducing perioperative opioid use, while improving the quality of surgical recovery when employing an Opioid Sparing Anesthesia (OSA) protocol with non-narcotic analgesics.

More than a million hernia repairs are performed each year in the US. With the significant nationwide obesity epidemic, it is estimated that the prevalence of hiatal hernias in the western population is approximately 20%. The investigators perform hundreds of laparoscopic hiatal hernia repairs annually at NorthShore University HealthSystem. Patients routinely receive fentanyl and other opioids during this surgery to reduce pain, but opioids also increase the risk of nausea, vomiting, and ileus. In addition, these patients are often times prescribed opioids upon discharge from the hospital. Preliminary results from a small, retrospective study among laparoscopic hiatal hernia surgical patients suggested that an OSA protocol with non-narcotic analgesics (that included dexmedetomidine and ketamine) resulted in a 33% reduction in those patients requiring opioids post-discharge. Moreover, these same patients had a significant reduction in hospital length of stay and nausea/retching. Therefore, the investigators propose a double-blinded randomized controlled trial to compare the number of patients in OSA protocol vs. Opioid Based Anesthesia (OBA) protocol groups, who require no opioids within 7 days postoperatively, (a time period where our quality data suggest nearly all patients receive postoperative opioids in this population).

ELIGIBILITY:
Inclusion Criteria:

* Patients from 18-90 years old who are undergoing laparoscopic hiatal hernia surgery
* Elective Laparoscopic hiatal hernia repair

Exclusion Criteria:

* Patients receiving urgent or emergent hiatal hernia surgery
* Patients receiving hiatal hernia surgery without laparoscopy
* Patients with adverse reactions (e.g., anaphylaxis, rash) to any of the drugs in the OBA or OSA protocols.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
The difference in discharge opioid consumption in morphine milligram equivalents (MMEs) | through postoperative Day 7
  The difference in discharge opioid consumption in morphine milligram equivalents (MMEs) through postoperative day 7 in patients in the Opioid Sparing Anesthesia (OSA) protocol vs. Opioid Based Anesthesia (OBA) protocol will be collected.

SECONDARY OUTCOMES:
Postoperative Visual Analogue Scale (VAS) pain scores | Upon post-anesthesia care unit arrival (within 2 hours after surgery), upon post-anesthesia care unit discharge (4 hours after surgery), and upon hospital discharge (up to 7 days)
  Patients Visual Analogue Scale (VAS) pain scores in each group will be collected. Subjects will rate their pain level on a scale of 0-10. Number "0" indicates no pain and number "10" indicates terrible pain.
Total Hospital Opioid Consumption (MMEs) | up to 7 days
  Total hospital opioid consumption (MMEs) in each group will be collected.
Post Anesthesia Care Unit | up to 7 days
  Post anesthesia care unit length of stay (hours) in each group will be recorded.
Hospital Length of stay | up to 7 days
  Hospital length of stay (days) in each group will be recorded.
Incidence of post operative nausea and vomiting (PONV ) | during post anesthesia care unit stay (up to 3 hours), postoperative Day 1, during hospital stay (up to 7 days)
  Incidence of post operative nausea and vomiting in each group will be recorded.
Rate of rehospitalization | within 30 days
  Rate of rehospitalization will be recorded for each group up to 30 days after hiatal hernia surgery.
Rate of reoperation | within 30 days
  Rate of reoperation will be recorded for each group up to 30 days after hiatal hernia surgery.
Rate of emergency room visit | within 30 days
  Rate of emergency room visits will be recorded up to 30 days after hiatal hernia surgery.
Surgeon satisfaction with surgical conditions | within 30 minutes after surgery
  Surgeon satisfaction with surgical conditions using a 5-point Likert score will be collected after surgery. A scale from 1-5; 1=Very dissatisfied, 2=Somewhat dissatisfied, 3=Neutral, 4=Somewhat satisfied, 5=Very satisfied)
Hospital Cost Differential | up to 30 days
  Hospital Cost Differential between groups while in hospital using direct operating cost.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Greenberg, MD, Principal Investigator — Endeavor Health
Locations (1):
- Endeavor Health, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lawal OD, Gold J, Murthy A, Ruchi R, Bavry E, Hume AL, Lewkowitz AK, Brothers T, Wen X. Rate and Risk Factors Associated With Prolonged Opioid Use After Surgery: A Systematic Review and Meta-analysis. JAMA Netw Open. 2020 Jun 1;3(6):e207367. doi: 10.1001/jamanetworkopen.2020.7367. PMID 32584407
- [Background] Bastawrous AL, Brockhaus KK, Chang MI, Milky G, Shih IF, Li Y, Cleary RK. A national database propensity score-matched comparison of minimally invasive and open colectomy for long-term opioid use. Surg Endosc. 2022 Jan;36(1):701-710. doi: 10.1007/s00464-021-08338-9. Epub 2021 Feb 10. PMID 33569727
- [Background] Siu EY, Moon TS. Opioid-free and opioid-sparing anesthesia. Int Anesthesiol Clin. 2020 Spring;58(2):34-41. doi: 10.1097/AIA.0000000000000270. No abstract available. PMID 32004171
- [Background] Bakan M, Umutoglu T, Topuz U, Uysal H, Bayram M, Kadioglu H, Salihoglu Z. Opioid-free total intravenous anesthesia with propofol, dexmedetomidine and lidocaine infusions for laparoscopic cholecystectomy: a prospective, randomized, double-blinded study. Braz J Anesthesiol. 2015 May-Jun;65(3):191-9. doi: 10.1016/j.bjane.2014.05.001. Epub 2014 Jun 3. PMID 25925031
- [Background] Hoffman C, Buddha M, Mai M, Sanjeevi S, Gutierrez R, O' Neill C, Miller A, Banki F. Opioid-Free Anesthesia and Same-Day Surgery Laparoscopic Hiatal Hernia Repair. J Am Coll Surg. 2022 Jul 1;235(1):86-98. doi: 10.1097/XCS.0000000000000229. Epub 2022 Apr 11. PMID 35703966
- [Background] Anderson R, Saiers JH, Abram S, Schlicht C. Accuracy in equianalgesic dosing. conversion dilemmas. J Pain Symptom Manage. 2001 May;21(5):397-406. doi: 10.1016/s0885-3924(01)00271-8. PMID 11369161
- [Background] Wengritzky R, Mettho T, Myles PS, Burke J, Kakos A. Development and validation of a postoperative nausea and vomiting intensity scale. Br J Anaesth. 2010 Feb;104(2):158-66. doi: 10.1093/bja/aep370. Epub 2009 Dec 26. PMID 20037151